CLINICAL TRIAL: NCT04653597
Title: Non-invasive Airway Management of Comatose Poisoned Emergency Patients
Acronym: NICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200013; 2020-A02036-33 (Other: ANSM)
Record Dates: First submitted 2020-10-09; First posted 2020-12-04 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Poisoning; Consciousness, Level Altered; Comatose
Keywords: ED; ICU; MICU; Coma; Comatose poisoning; intubation; Endotracheal intubation; GCS; Glasgow Coma Scale
MeSH Terms: conditions — Poisoning; Consciousness Disorders; Coma | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative airway management (Experimental): decision to intubate will be withheld as long as the patient's state allows it. The patient will be closely monitored and decision of intubation will be made upon presence of regurgitation, seizure, shock, or sign of respiratory distress.
  Interventions: Procedure: Close monitoring
- Routine practice (Other): decision of intubation left at the discretion of the emergency physician
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Close monitoring — surveillance every 30 minutes of blood pressure, SpO2, respiratory rate, heart rate and GCS until the patient recovers a GCS>8 or responds adequately to a simple order
  Arms: Conservative airway management
Procedure: Endotracheal intubation — invasive airway management in order to avoid risk of pulmonary aspiration
  Arms: Routine practice

SUMMARY:
A decreased level of consciousness is a common reason for presentation to the emergency department (ED) and is often the result of intoxication (up to 1% of all ED visits and 3% of ICU admission). In France, approximately 165 000 poisoned patients are managed each year. Originally developed in head injured patients, the Glasgow Coma Scale (GCS) is a validated reproducible score evaluating the level of consciousness: a GCS ≤ 8 is strongly associated with reduced gag reflex and increased incidence of aspiration pneumonia. Although recommended for patients with traumatic brain injury and coma, it remains unknown whether the benefit of an invasive management of airways with sedation, intubation and mechanical ventilation should be applied to other causes of coma in particular for acute poisoned patients. The investigator hypothesize that a conservative management with close monitoring without immediate endotracheal intubation of these patients is effective and associated with less in-hospital complications (truncated at 28 days) compared to routine practice management (in which the decision of immediate intubation is left to the discretion of the emergency physician).

DETAILED DESCRIPTION:
A decreased level of consciousness is a common reason for presentation to the emergency department (ED) and is often the result of intoxication (up to 1% of all ED visits and 3% of intensive care unit (ICU) admission). In France, approximately 165 000 poisoned patients are managed each year.1 Originally developed in head injured patients, the Glasgow Coma Scale (GCS) is a validated reproducible score evaluating the level of consciousness - a GCS ≤ 8 is associated with reduced gag reflex and increased incidence of aspiration pneumonia (with an adjusted odds ratio of 2.32, 95%CI =1.60 to 3.33). However, whether this risk of aspiration pneumonia (AP) may be decreased by early intubation is unknown, and no difference in the risk of AP was reported between patients that were intubated early and patients who were not.

Although it is well established that in trauma patients, a GCS ≤ 8 mandates airway management by endotracheal intubation, it remains unknown whether this strategy should be applied to other etiologies of coma, in particular for acute poisoned patients. Tracheal intubation and mechanical ventilation allow to prevent aspiration pneumonia, to optimize oxygenation and gas exchange.

Investigators will include patients with a decreased level of consciousness (defined by a GCS of 8 or less) caused by acute intoxication (alcohol, recreative drugs, or other prescription drugs (with the exception intoxication with cardiotropic drugs, e.g. beta blockers, calcium channel inhibitor, angiotensin conversion enzyme)). These patients will be included at the initial stage of their management: in the ED, or out of hospital with a pre-hospital emergency physician. Patients with clear proven benefit of intubation will be excluded : patients in shock, patients with suspicion of brain lesion, seizure related with poisoning, visualization of regurgitation of gastric content or sign of respiratory distress. Conservative airway management. Patients will be conservatively managed, i.e. close monitoring and no intubation and mechanical ventilation unless the patient presents a clinical event that needs intubation (shock, sign of respiratory distress, visualization of regurgitation or seizure).

Acute poisoning is a common reason for presentation to the ED or MICU intervention (up to 1% of all ED visits and 3% of intensive care unit (ICU) admission). These patients are often intubated (reported rate ranging from 20 to 50% in different cohort studies), when their GCS is below 8, in order to protect their airways. However there is currently no clear demonstration of its efficacy in this specific target population, while it is known that intubation is associated with morbidity and mortality.

Intubated patients need subsequent intensive care unit admission and invasive monitoring, and this can be associated with increased risk of pulmonary complications, length of hospital-stay, nosocomial infections and cost. In a context of expenditures control in health care, appropriate intensive care resource utilization is an important issue. When considering the increasing demand for intensive care among emergency patients, the importance of health care resource allocation and expenditure control, and the possible absence benefit of intubation and intensive care, an endotracheal airway management of poisoned coma patients might be detrimental.

Thus, if our hypothesis is demonstrated, the results of NICO study will change practice and guidelines for management of acute coma poisoned patients, with less exposure to the morbidity of endotracheal intubation and associated with decrease of ICU stay, and reduction of their health costs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Clinical suspicion of acute poisoning (either alcohol, drug or medication)
3. Decreased level of consciousness with a GCS ≤ 8 assessed by an emergency physician either in the ED or in the out of hospital field with the mobile intensive care unit (MICU).
4. Written informed consent signed by the patient / the trustworthy person / family member / close relative or inclusion in case of emergency
5. Patients affiliated to French social security ("AME" excepted)

Exclusion Criteria:

1. Respiratory failure (SpO2 < 90% with oxygen provided by nasal cannula (≤ 4 l/min.), clinical signs of respiratory distress)
2. Sustained systolic blood pressure < 90 mmHg despite fluid resuscitation of 1 liter of critalloid
3. Witnessed seizure
4. Acute cerebral aggression (Traumatic brain injury, intracranial hematoma, stroke)
5. Suspected Cardiotropic drugs poisoning (beta blockers, calcium channel inhibitor, angiotensin conversion enzyme), QRS or QT enlargement on ECG.
6. Suspected sole intoxication with toxic for which there is an antidote
7. Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom
8. Known Pregnant women and breast feeding woman
9. Participation in another intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Hierarchical composite endpoint of (truncated at 28 days): - In hospital death | at 28 days
  this endpoint will be reported using both the Finkelstein model (Finkelstein Stat med 1999; Beitler JAMA 2019) and the win ratio methods (Pocok Eur H J 2016), with priority listed in this order from highest to lowest. Patients will be followed until hospital discharge (or truncated at 28 days if still hospitalized) and data collected in the electronic health record the investigator with the help of a clinical research technician.
Hierarchical composite endpoint of (truncated at 28 days):- Length of ICU stay | at 28 days
  this endpoint will be reported using both the Finkelstein model (Finkelstein Stat med 1999; Beitler JAMA 2019) and the win ratio methods (Pocok Eur H J 2016), with priority listed in this order from highest to lowest. Patients will be followed until hospital discharge (or truncated at 28 days if still hospitalized) and data collected in the electronic health record the investigator with the help of a clinical research technician.
Hierarchical composite endpoint of (truncated at 28 days): - Length of hospital stay | at 28 days
  this endpoint will be reported using both the Finkelstein model (Finkelstein Stat med 1999; Beitler JAMA 2019) and the win ratio methods (Pocok Eur H J 2016), with priority listed in this order from highest to lowest. Patients will be followed until hospital discharge (or truncated at 28 days if still hospitalized) and data collected in the electronic health record the investigator with the help of a clinical research technician.

SECONDARY OUTCOMES:
In-hospital death (truncated at 28 days) | at 28 days
  number of included patients dead at 28 days after randomisation
ICU length of stay (truncated at 28 days) | at 28 days
  number of day in ICU for each patient included since randomization
Hospital length of stay (truncated at 28 days) | at 28 days
  number of day in hospitalization for each patient included since their randomization
Proportion of patient with Mechanical ventilation at day 28 | at 28 days
  number of patient included with mechanical ventilation 28 days after randomization
Lenght of mechanical ventilation until hospital discharge or at day28 | at 28 days
Proportion of ICU admission | 28 days
  number of patient included admitted to ICU during hospital stay
Proportion of rapid onset pneumonia | 28 days
  number of patient included developing a rapid onset pneumonia during hospital stay
Adverse events from intubation (hypoxemia, dental trauma, regurgitation, cardiac arrest, intubation difficulty score (IDS) ≥ 5, hypotension or esophageal intubation) | 28 days
  number of patient included developing an adverse events from intubation during hospital stay, and type of adverse events
total hospital costs (truncated at 28 days) | at 28 days
  cost of hospitalization for patient included in the study.
total hospital cost consequence analysis (truncated at 28 days) | at 28 days
  cost of hospitalization for patient included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan FREUND, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siaha BFN, Ossima AN, Mimouni M, Freund Y, Durand-Zaleski I; NICO Study Group. Cost-effectiveness of non-invasive airway management of comatose patients with acute poisoning. Intensive Care Med. 2024 Jul;50(7):1169-1171. doi: 10.1007/s00134-024-07452-1. Epub 2024 Jun 24. No abstract available. PMID 38913094
- [Derived] Freund Y, Viglino D, Cachanado M, Cassard C, Montassier E, Douay B, Guenezan J, Le Borgne P, Yordanov Y, Severin A, Roussel M, Daniel M, Marteau A, Peschanski N, Teissandier D, Macrez R, Morere J, Chouihed T, Roux D, Adnet F, Bloom B, Chauvin A, Simon T. Effect of Noninvasive Airway Management of Comatose Patients With Acute Poisoning: A Randomized Clinical Trial. JAMA. 2023 Dec 19;330(23):2267-2274. doi: 10.1001/jama.2023.24391. PMID 38019968